CLINICAL TRIAL: NCT04993716
Title: Epidemiological Study on the Management of Out-of-hospital Cardiac Arrest Survivors in Champagne ArDEnnes
Acronym: CASCADE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Stephane Sanchez (Other)
Responsible Party: Sponsor-Investigator, Stephane Sanchez, Sponsor, Centre Hospitalier de Troyes
Organization: Centre Hospitalier de Troyes (Other)
Other Study IDs: The CASCADE Study
Record Dates: First submitted 2021-06-18; First posted 2021-08-06 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Out-of-hospital Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: Patient present in the SAU after an extra-hospital cardiac arrest
  Interventions: Other: observational

INTERVENTIONS:
Other: observational — Collect from a bank of biological samples, identification of prognostic factors associated with survival without serious neurological heavy sequelae

SUMMARY:
Out-of-hospital cardiac arrest (OHCA) is a public health problem, affecting 50,000 people per year in France. Intervention time (initiation of cardiopulmonary resuscitation (CPR) and advanced CPR) are associated with a better prognosis. Despite this, the latest published data show a very low overall survival (5%). Our territory has only three centers distributed hospitals with both a 24-hour coronary angiography platform and an intensive care unit. Finally, although 60% of ACEHs receive coronary angiography in the Île de France region, it is performed on only 15% of patients in the Reims University Hospital.

Therefore, it seems essential to conduct a study on the reality of the support of ACEH and to study the clinical and biological factors as well as the influence of the geographical distribution of specialized technical platforms on the prognosis of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient victim of ACEH in the Champagne-Ardenne region admitted living in hospital.

Exclusion Criteria:

* patient under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our participants must be the victim of an ACEH on the Champagne-Ardenne territory admitted living in the hospital and be over eighteen years old
Sampling Method: Non-Probability Sample
Enrollment: 294 (Estimated)
Dates: Start 2021-10-04 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Analysis of prognostic factors associated with survival without severe neurological sequelae (CPC 1-2) at 3 months among the following variables | 3 months
Analysis of prognostic factors associated with survival without severe neurological sequelae (CPC 1-2) with collection of a bank of biological samples, identification of clinical factors and targeted temperature control | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- hospital center of Troyes, Troyes, Champagne Ardennes, France

IPD SHARING:
Plan to Share IPD: No